CLINICAL TRIAL: NCT04097262
Title: Price Elasticity of Fruit (Shop For Success)
Brief Title: Shop For Success: Experimental Grocery Store Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Grand Forks Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: GFHNRC155
Record Dates: First submitted 2019-09-18; First posted 2019-09-20 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: This study will utilize a three factor design, with one between-subject factor and two within-subject factors. The between-subject factor is participation in a federal food assistance program. The within-subject factors are price change condition and price change scenario.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Own-Price Elasticity (Experimental): The price of fruit will vary (own-price elasticity) while the price of all other foods in the "mock" grocery store will remain constant.
  Interventions: Other: Own-Price Elasticity
- Cross-Price Elasticity (Experimental): The price of fruit will remain constant while the price of other foods in the "mock" grocery store will vary (cross-price elasticity).
  Interventions: Other: Cross-Price Elasticity

INTERVENTIONS:
Other: Own-Price Elasticity — The price of fruit will be 75%, 100%, or 125% of the reference price, but the price of other foods will remain the same.
  Arms: Own-Price Elasticity
Other: Cross-Price Elasticity — The price of fruit will remain the same, but the price of other foods will be 75%, 100%, or 125% of the reference price.
  Arms: Cross-Price Elasticity

SUMMARY:
The purpose of this research is to study how the price of foods affects food buying choices at the grocery store. The researchers are interested in this topic because the price of foods can have a big impact on what people choose to buy and prices change over time. The researchers are doing this study to see how changes in food prices affect what foods mothers choose for their families.

DETAILED DESCRIPTION:
It is well known that the price of a given food affects the amount of that food an individual purchases. However, little is known about how specific groups, such as overweight/obese and those with lower incomes, change their food purchasing decisions depending on food price changes. Evidence has shown that these groups have lower quality diets and worse health outcomes than their normal weight and higher income counterparts. Therefore, it is important to gain a better understanding of how food price changes affect purchasing decisions among these populations in order to develop targeted nutrition interventions to improve their diet quality. To investigate this, the researchers will create a laboratory-based grocery store, in which pictures of foods will be used to substitute actual food. Food prices will be indicated on each picture. Participants will be given play money and a budget, and ask them to "purchase" foods in the mock grocery store. The price of food will be changed throughout the study to investigate how participants change their purchasing decisions based on these price changes.

ELIGIBILITY:
Inclusion Criteria:

* Have at least one child up to 18 years of age residing in the household
* Primary grocery shopper for the household
* No health conditions or food practices that substantially limit food choice
* Not currently pregnant
* Consent to the study design

Exclusion Criteria:

* Male
* < 18 years of age
* Not a mother, or children not living with subject in their household
* No children below the age of 18 years of age
* Not the primary grocery shopper for their household
* Health conditions or food practices that substantially limit food choice
* Currently pregnant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2019-08-22 (Actual); Primary Completion 2020-03-25 (Actual); Study Completion 2020-03-25 (Actual)

PRIMARY OUTCOMES:
Price elasticity of fruit | Baseline
  Percent change in the amount of fruit purchased (gram weight) for every percent change in the price of a given food.

SECONDARY OUTCOMES:
Nutrient density of purchased foods | Baseline
  Ratio of low nutrient-dense food purchases to high nutrient-dense food purchases

CONTACTS AND LOCATIONS:
Overall Officials: James Roemmich, PhD, Principal Investigator — USDA Grand Forks Human Nutrition Research Center
Locations (1):
- USDA Grand Forks Human Nutrition Research Center, Grand Forks, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2019-08-16): https://cdn.clinicaltrials.gov/large-docs/62/NCT04097262/ICF_000.pdf